CLINICAL TRIAL: NCT04428827
Title: Long-term Outcomes in Patients With Primary Aldosteronism After Treatment
Brief Title: Outcome of Patients With Primary Aldosteronism
Acronym: PA_Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PA_Outcome
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Primary Aldosteronism; Primary Aldosteronism Due to Aldosterone Producing Adenoma; Primary Aldosteronism Due to Adrenal Hyperplasia (Bilateral); Adrenalectomy; Status; Mineralocorticoid Excess; Mineralocorticoid Antagonists [Aldosterone Antagonists] Causing Adverse Effects in Therapeutic Use; Cardiovascular Morbidity; Chronic Renal Disease; Hypokalemia
MeSH Terms: conditions — Hyperaldosteronism; Renal Insufficiency, Chronic; Hypokalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery: Patients treated with surgery
  Interventions: Procedure: Unilateral adrenalectomy in patients with unilateral disease
- Medications: Patients treated with mineralocorticoid antagonists or potassium sparing diuretics for primary aldosteronism

INTERVENTIONS:
Procedure: Unilateral adrenalectomy in patients with unilateral disease — Unilateral adrenalectomy in patients with unilateral disease
  Groups: Surgery

SUMMARY:
Majority of patients with hypertension have primary hypertension (without an underlying cause). Primary aldosteronism (PA) is the most common cause of secondary hypertension, and can be found in 5-10% of patients locally. PA is caused by excessive release of a hormone (aldosterone) from the adrenal glands, which can be unilateral (one gland) or bilateral (both glands).

It has been shown that excess aldosterone has other harmful effects in addition to hypertension, such as directly affecting the heart, blood vessels, kidneys, leading to increased cardiovascular morbidity and mortality. This is supported by studies showing reversal of these effects after treatment for PA.

The investigators aim to assess the long-term cardiovascular, and renal outcomes of patients with PA, compared to patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected primary aldosteronism

Exclusion Criteria:

* Nil

Ages: 14 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected primary aldosteronism managed at referral centre for suspected primary aldosteronism
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
change in systolic blood pressure before and after treatment | six months after treatment
  change in systolic blood pressure

SECONDARY OUTCOMES:
change in diastolic blood pressure before and after treatment | six months after treatment
  change in diastolic blood pressure
change in systolic blood pressure before and after treatment | through study completion, an average of 5 years
  change in systolic blood pressure
change in diastolic blood pressure before and after treatment | through study completion, an average of 5 years
  change in diastolic blood pressure
cardiovascular outcome | through study completion, an average of 5 years
  incidence of new cardiovascular events including acute myocardial infarction, revascularisation percutaneously, coronary artery bypass graft, stroke, admission for congestive cardiac failure, atrial fibrillation
chronic kidney disease | through study completion, an average of 5 years
  incidence of worsening chronic kidney disease, decline of glomerular filtration rate by 15ml/min from at least 60m/min
Renal Progression | through study completion, an average of 5 years
  rate of decline of glomerular filtration rate
variables that predict unilateral disease | through study completion, an average of 5 years
  Identify variables that are more common in patients with unilateral disease
variables that predict blood pressure response | through study completion, an average of 5 years
  Identify variables that are more common in patients with positive blood pressure response

CONTACTS AND LOCATIONS:
Overall Officials: Troy Puar, MRCP, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of anonymised pooled data

REFERENCES:
- [Derived] Puar TH, Loh LM, Loh WJ, Lim DST, Zhang M, Tan PT, Lee L, Swee DS, Khoo J, Tay D, Tan SY, Zhu L, Gani L, King TF, Kek PC, Foo RS. Outcomes in unilateral primary aldosteronism after surgical or medical therapy. Clin Endocrinol (Oxf). 2021 Feb;94(2):158-167. doi: 10.1111/cen.14351. Epub 2020 Oct 26. PMID 33058182